CLINICAL TRIAL: NCT04889417
Title: COgnitive and Physical Exercise to Improve Outcomes After Surgery (COPE-iOS) Study
Acronym: COPEiOS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Christopher G Hughes, Professor of Anesthesiology, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: U11775; 1R01AG061161-01A1 (NIH)
Record Dates: First submitted 2021-04-01; First posted 2021-05-17 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Cognitive Impairment; Disability Physical; Surgery
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Treatment assignment will be known only by the research coordinators, therapists, and research staff overseeing the administration of the program or active control. The remaining research staff, neuropsychology professionals performing the assessments, and clinicians will be blinded. Participants will be blinded to their group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Computerized brain game training and online interactive physical exercise training
  Interventions: Behavioral: Comprehensive training program
- Control (Active Comparator): Control computer games and online interactive stretching exercises.
  Interventions: Behavioral: Active control

INTERVENTIONS:
Behavioral: Comprehensive training program — The COPE-iOS program is a pragmatic comprehensive training program that combines computerized cognitive training and progressive supervised video conference physical exercise sessions performed 2-4 weeks prior to surgery and for 3 months after discharge.
  Arms: Intervention
Behavioral: Active control — The active attention control will include control computer games and supervised video conference stretching exercises performed 2-4 weeks prior to surgery and for 3 months after discharge.
  Arms: Control

SUMMARY:
The COgnitive and Physical Exercise to improve Outcomes after Surgery (COPE-iOS) study is testing the hypothesis that a pragmatic program combining computerized cognitive training and physical training throughout the perioperative period will improve long-term cognitive and disability outcomes in older surgical patients at high risk for decline. To accomplish these goals, the Investigators are randomizing 250 patients ≥60 years old undergoing elective major non-cardiac surgery with expected hospitalization ≥3 days to a pragmatic comprehensive training program (computerized cognitive training and supervised progressive physical exercise) or to active control (control computer game, stretching exercises) for 2-4 weeks prior to surgery and for 3 months after discharge. At baseline and after discharge, the Investigators will assess global cognition, activities of daily living, depression, endothelial and blood brain barrier function (blood biomarkers), and neuroimaging (anatomical and functional MRI). In this early stage trial, the Investigators will determine if certain subgroups benefit most, program aspects with greatest effect on outcomes, mechanistic associations with outcomes, and additional exploratory analyses.

ELIGIBILITY:
Inclusion Criteria:

1. ≥60 years old
2. undergoing elective major non-cardiac surgery with expected hospitalization ≥3 days

Exclusion Criteria:

1. Blind, deaf, or inability to understand English as these conditions would preclude the ability to perform the proposed comprehensive program and prevent assessment with the study instruments
2. Prisoners
3. Severe frailty or physical impairment that prohibits participation in the program
4. Cognitively unable to consent for surgery (i.e., dementia or cognitive impairment of a severity that precludes ability to self-consent and, thus, also participation in study interventions)
5. Inability to obtain informed consent ≥2 weeks before scheduled surgery
6. Surgical team unwilling to allow physical activity or other components of the intervention
7. Inability or unwillingness to utilize a tablet device, laptop, or email
8. Co-enrolled in another interventional trial examining similar outcomes or current enrollment in a study that does not allow co-enrollment

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Global cognition | 3 months after discharge
  Computerized Neuropsychological Scale (CNS) Vital Signs neurocognitive battery

SECONDARY OUTCOMES:
Global cognition | 12 months after discharge
  Computerized Neuropsychological Scale (CNS) Vital Signs neurocognitive battery
Basic activities of daily living | 3 and 12 months after discharge
  Katz activities of daily living
Instrumental activities of daily living | 3 and 12 months after discharge
  Functional activities questionnaire
Depression | 3 and 12 months after discharge
  Depression Anxiety and Stress Scale (DASS)
Endothelial injury | day of surgery, postoperative day 2, postoperative day 5, and 3 months after discharge
  Plasma biomarker
Blood brain barrier injury | day of surgery, postoperative day 2, postoperative day 5, and 3 months after discharge
  Plasma biomarker
Brain magnetic resonance imaging | 3 months after discharge
  Anatomical and functional magnetic resonance imaging of the brain

OTHER OUTCOMES:
Program compliance | before surgery up to 3 months after discharge
  Compliance with program, feasibility, including sessions attended and completed, heart rate and exertion tracking during session
Delirium | up to 14 days in the hospital
  Confusion assessment method in the ICU
Length of stay | through hospital admission, an average of up to 14 days
  Length of stay in the hospital
Discharge location | through hospital admission, an average of up to 14 days
  Home, rehabilitation, skilled nursing facility, hospice
Functional status | 3 and 12 months after discharge
  Duke Activity Status Index
Chronic Pain | 3 and 12 months after discharge
  Behavioral Pain Index
Adverse events | before surgery up to 3 months after discharge
  Safety evaluated by adverse event monitoring, including physical injury (e.g., discomfort, falls, myocardial ischemia, syncope, dyspnea), above maximum heart rate, and fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G Hughes, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes